CLINICAL TRIAL: NCT01459874
Title: Prospective Registry for the Evaluation of an Organizational Model for Remote Monitoring of Pacemaker and Implantable Cardioverter Defibrillator (ICD) Recipients in the Clinical Practice
Brief Title: Evaluation of an Organizational Model for Remote Monitoring of Pacemaker and Implantable Cardioverter Defibrillator Recipients
Status: Completed | Type: Observational
Sponsor: San Filippo Neri General Hospital (Other)
Collaborators: Biotronik Italia (Industry)
Responsible Party: Principal Investigator, Renato Pietro Ricci, Principal Investigator, San Filippo Neri General Hospital
Other Study IDs: HomeGuide
Record Dates: First submitted 2011-10-24; First posted 2011-10-26 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Pacemaker; Implantable Cardioverter Defibrillator
Keywords: Home Monitoring; Remote monitoring; Telecardiology; Organizational model; Patient indicated for pacemaker, ICD, CRT-P, or CRT-D
MeSH Terms: interventions — Models, Organizational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cardiac Implantable Device recipients
  Interventions: Behavioral: Organizational model for remote monitoring

INTERVENTIONS:
Behavioral: Organizational model for remote monitoring — An organizational model defining roles and behaviors of subjects involved in the remote monitoring of pacemaker and defibrillator recipients
  Other Names: Biotronik Home Monitoring

SUMMARY:
The purpose of the registry is to evaluate an organizational model fixing roles and behaviors of subjects involved in the remote monitoring of patients implanted with pacemakers and defibrillators.

The evaluation will estimate the clinical efficiency and the impact on health service resources of the organizational model when this is implemented in the daily clinical practice.

DETAILED DESCRIPTION:
After a number of studies which assessed technical reliability and clinical implications of remote monitoring systems, a further step should approach the issue of how remote monitoring can be implemented as a part of routine activities of a cardiology outpatient clinic. A clear definition of roles and workflow to timely manage information and properly react to adverse events is required. The HomeGuide Registry proposes an organizational model specifying roles and procedures for outpatient clinics using a specific remote monitoring system in routine follow-up. The HomeGuide model is essentially based on an interaction between one or more allied professionals (expert and trained nurses or technicians) and a responsible physician. The main objective of the HomeGuide Registry is to evaluate:

1. Clinical efficiency of remote patient management;
2. Health service resources required by a remote patient management.

ELIGIBILITY:
Inclusion Criteria:

* Patients implanted with a BIOTRONIK pacemaker or ICD with Home Monitoring (HM) technology
* Ability to utilize the HM system throughout the study
* Ability to give informed consent
* Ability to return for regular follow-ups for two years

Exclusion Criteria:

* Patients who do not fulfill all inclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Cardiac Implantable Device recipients
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Actual)
Dates: Start 2008-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity, positive predictive value and expected utility of the organizational model | Up to two years
  Sensitivity, positive predictive value and expected utility in the detection of all cardiovascular and device-related events of the proposed organizational model

SECONDARY OUTCOMES:
Manpower of the organizational model | Up to two years
  Health care source consumption required to implement the organizational model for the remote management of patients

CONTACTS AND LOCATIONS:
Overall Officials: Renato Pietro Ricci, Principal Investigator — San Filippo Neri Hospital, Rome, Italy; Loredana Morichelli, Study Chair — San Filippo Neri Hospital, Rome, Italy; Gianfranco Buja, Study Chair — Policlinico universitario, University of Padua, Italy; Leonardo Calò, Study Chair — Policlinico Casilino, Rome, Italy; Antonio Curnis, Study Chair — Spedali Civili, University of Brescia, Italy; Antonio D'Onofrio, Study Chair — Monaldi Hospital, Italy; Diego Vaccari, Study Chair — Montebelluna Hospital, Italy; Gabriele Zanotto, Study Chair — Legnago Hospital, Verona, Italy; Alessio Gargaro, Study Chair — Biotronik Italia; Nicola Rovai, Study Chair — Biotronik Italia
Locations (74):
- Italy (74):
  - Senigallia Civil Hospital, Senigallia, Ancona
  - Presidio Ospedale di Ariano Irpino, Ariano Irpino, Avellino
  - Umberto I Hospital, Altamura, Bari
  - Michele Sarcone Hospital, Terlizzi, Bari
  - PO Francesco Ferrari, Casarano, Lecce
  - P.O.G. Fogliani, Milazzo, Messina
  - Ospedale di Circolo, Desio, Monza E Brianza
  - San Leonardo, Castellammare di Stabia, Napoli
  - Volterra Hospital, Volterra, Pisa
  - SS. Cosimo e Damiano Hospital, Pescia, Pistoia
  - P. O. Villa D'Agri, Marsicovetere, Potenza
  - Guizzardi Hospital, Vittoria, Ragusa
  - G. B. Grassi, Ostia Antica, Roma
  - Santa Maria Della Misericordia Hospital, Sorrento, Salerno
  - P.O. Giannuzzi, Manduria, Taranto
  - Paolo Borsellino Hospital, Marsala, Trapani
  - Ulss n. 7, Conegliano, Treviso
  - Montebelluna Hospital, Montebelluna, Treviso
  - ULSS n. 14, Chioggia, Venezia
  - Dell'Angelo Hospital, Mestre, Venezia
  - Mirano Hospital, Mirano, Venezia
  - Portogruaro Hospital, Portogruaro, Venezia
  - Mater Salutis Hospital, Legnago, Verona
  - G.M. Lancisi Hospital, Ancona
  - I.N.R.C.A., Ancona
  - S. Donato di Arezzo Hospital, Arezzo
  - Policlinico - Card. Universitaria, Bari
  - Policlinico - Cardiologia Ospedaliera, Bari
  - Policlinico - Cardiologia Ospedaliera, Benevento
  - AO Spedali Civili, Brescia
  - Congreg. Ancelle della Carità Poliambulanza, Brescia
  - A. Perrino Hospital, Brindisi
  - Cardarelli Hospital, Campobasso
  - S. Cuore University, Campobasso
  - Carrara Civil Hospital, Carrara
  - Sant'Anna e San Sebastiani Hospital, Caserta
  - Ferrarotto Hospital, Catania
  - AO Arcispedale S. Anna, Ferrara
  - A.O.U. Careggi S.O.D. Aritmologia, Florence
  - S. Giovanni di Dio Hospital, Florence
  - S. Maria Annunziata Hospital, Florence
  - S. Maria Nuova Hospital, Florence
  - P.O. Di Gorizia, Gorizia
  - F. Veneziale Hospital, Isernia
  - Vito Fazzi Hospital, Lecce
  - Piemonte Hospital, Messina
  - Sacco Hospital, Milan
  - F.B.F., Napoli
  - Federico II Hospital, Napoli
  - Monaldi Hospital - Gruppo Sun, Napoli
  - Monaldi Hospital, U.O. Aritmologia, Napoli
  - Policlinico Federico II, Napoli
  - Policlinico Universitario di Padova, Padua
  - ARNAS Civico, Palermo
  - Cervello Hospital, Palermo
  - Santa Maria della Misericordia Hospital, Perugia
  - Guglielmo da Saliceto Civil Hospital, Piacenza
  - Santa Maria degli Angeli Hospital, Pordenone
  - Santa Maria Nuova Hospital, Reggio Emilia
  - Degli Infermi Hospital, Rimini
  - Casa di Cura Villa Pia, Roma
  - Policlinico Casilino, Roma
  - Policlinico Tor Vergata, Roma
  - Policlinico Umberto I, Roma
  - San Filippo Neri Hospital, Rome
  - San Giovanni di Dio e Ruggi D'Aragona Hospital, Salerno
  - San Donà di Piave Hospital, San Donà di Piave
  - Teresa Masselli Mascia Hospital, San Severo
  - P.O. SS. Annunziata, Taranto
  - Sant'Antonio Abate Hospital, Trapani
  - Ca' Foncello Hospital, Treviso
  - Di Circolo Hospital, Varese
  - Macchi Hospital, Varese
  - SS. Giovanni e Paolo Hospital, Venezia

REFERENCES:
- [Result] Ricci RP, Morichelli L, D'Onofrio A, Calo L, Vaccari D, Zanotto G, Curnis A, Buja G, Rovai N, Gargaro A. Effectiveness of remote monitoring of CIEDs in detection and treatment of clinical and device-related cardiovascular events in daily practice: the HomeGuide Registry. Europace. 2013 Jul;15(7):970-7. doi: 10.1093/europace/eus440. Epub 2013 Jan 29. PMID 23362021